CLINICAL TRIAL: NCT04344678
Title: The Phosphodiesterase 5 Inhibitor Sildenafil as an Adjunct to Antidepressants in Major Depressive Disorder Patients: Randomized, Double-Blind, Placebo-Controlled Trial
Brief Title: The Phosphodiesterase 5 Inhibitor Sildenafil as an Adjunct to Antidepressants in Major Depressive Disorder Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Institutional and funding constrains
Sponsor: Sadat City University (Other)
Responsible Party: Principal Investigator, Mahmoud Samy Abdallah, Lecturer of Clinical Pharmacy, PhD., Sadat City University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0044/2020
Record Dates: First submitted 2020-04-09; First posted 2020-04-14 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Sildenafil Citrate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Placebo Comparator): Escitalopram 20 mg tablet plus one placebo tablet
  Interventions: Drug: Placebo oral tablet
- Sildenafil group (Experimental): Escitalopram 20 mg tablet plus one Sildenafil 50 mg tablet
  Interventions: Drug: Sildenafil Citrate

INTERVENTIONS:
Drug: Sildenafil Citrate — Esitalopram 20 mg tablet plus Sildenafil Citrate 50 mg tablet once daily
  Arms: Sildenafil group
Drug: Placebo oral tablet — Esitalopram 20 mg tablet plus placebo tablet once daily
  Arms: Control group

SUMMARY:
Antidepressant-like effects of sildenafil to its ability to modulate transduction pathways responsible for neuroplasticity. Treatment with sildenafil was shown to be PKG-dependent and lead to increased expression of cGMP, pCREB, BDNF and VGF in the hippocampus and prefrontal cortex (PFC), brain areas relevant to mood disorders pathophysiology. Sildenafil produces antidepressant-like effects by inhibiting oxidative stress in the hippocampus and by decreasing the levels of IL-1β in the hippocampus and striatum.

ELIGIBILITY:
Inclusion Criteria:

* Eighty adult outpatients with the Diagnostic and Statistical Manual of Mental Disorders-IV (DSM-IV) diagnosis of MDD based on a MINI Neuropsychiatric Interview (MINI) (American Psychiatric Association., 2000; Sheehan et al., 1998), without psychotic features and a total 17 item HAM-D score of at least 18 with item 1 (depressed mood) scored 2 or greater were eligible (Hamilton, 1960).
* Patients were requested to be free of all the psychotropic and anti-inflammatory medications for at least 4 weeks before participating in the study.

Exclusion Criteria:

* Patients with bipolar I or bipolar II disorder
* Patients with personality disorders
* Patients with eating disorders
* Patients with substance dependence or abuse
* Patients with concurrent active medical condition
* Patients with history of seizures
* Patients with history of receiving Electroconvulsive therapy (ECT)
* Patients with inflammatory disorders
* Patients with allergy or contraindications to the used medications
* Patients with finally pregnant or lactating females
* Cardiovascular disorders
* Severe renal impairment: creatinine clearance of ≤ 25 ml/min
* Moderate or severe hepatic impairment

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Effect on Hamilton Depression rating scale score (HAM-D score) | 12 week
  The principal measure of the outcome was the 17-items HAM-D. Scoring is based on the 17-item scale and scores of 0-7 are considered as being normal, 8-13 suggest mild depression, 14-17 moderate depression and scores over 17 are indicative of severe depression. Remission is defined as HAM-D total score ≤ 7 (primary outcome). Treatment response is defined as ≥ 50% drop in the HAM-D total score.

SECONDARY OUTCOMES:
Effect on biological markers | 12 week
  Serum level of tumor necrosis factor alpha (TNF-α), Interleukin-6 (IL-6), and brain derived neurotrophic factor (BDNF) were measured at the baseline and after the treatment to evaluate the biological effects of the used medications.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Shibīn al Kawm, Egypt